CLINICAL TRIAL: NCT06216743
Title: PRE- MISTIC: MRI and Cine Imaging to Improve Staging of Tumors in the Colon
Acronym: PRE-MISTIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 84414
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-01

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Imaging cohort (Experimental): Patients participating in pilot study who will receive an additional MRI-scan, cineMRI and cineCT scan.
  Interventions: Diagnostic Test: MRI and CT

INTERVENTIONS:
Diagnostic Test: MRI and CT — Patients will undergo an additional MRI, cineMRI and CineCT cscan.

SUMMARY:
At this moment, we use CT and endoscopy to clinically stage colon tumours. Unfortunately, the combination of these imaging techniques is highly inaccurate. 40% of advanced pathological colon tumours (so called T4 tumours) are not staged as a T4 tumour pre-operatively. Preoperative or neoadjuvant chemotherapy (NAC) has improved outcomes in other gastrointestinal cancers and seems to be a promising pretreatment for colon tumours. To implement NACin colon tumours, we first need to stage the colon tumours with much higher accuracy. MRI sequences and cine imaging hold promise to provide more accurate staging of colon tumours.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical suspicion for T3 or T4 tumor based on standard clinical work-up with endoscopy and CT-scan
* Age > 18 years
* WHO Performance status of 0-2

Exclusion Criteria:

* Patients with contraindications for MRI
* Patients with clinical contraindications to undergo colon surgery
* Patients receiving neoadjuvant therapy prior to surgery
* Patients with known allergy to iodine or gadolinium contrast
* Patient with contra-indication for contrasts based on kidney failure Neoadjuvant therapy is currently not the standard of care for advanced colon carcinoma, and applied only in selected cases or as part of a clinical trial. Because neoadjuvant therapy could result in tumor regression, thus impacting the gold standard of histological examination, patients selected for neoadjuvant therapy are excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of different MRI sequences to diagnose T4 colon carcinoma. | 6 weeks

SECONDARY OUTCOMES:
Sensitivity and specificity of different MRI sequences, including diffusion weighted imaging, to diagnose N2 disease, as compared to the golden standard of histological examination. | 6 weeks
Establishing an MRI Protocol that is optimized for the clinical staging of colon tumors | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Nijmegen Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Morton D, Seymour M, Magill L, Handley K, Glasbey J, Glimelius B, Palmer A, Seligmann J, Laurberg S, Murakami K, West N, Quirke P, Gray R; FOxTROT Collaborative Group. Preoperative Chemotherapy for Operable Colon Cancer: Mature Results of an International Randomized Controlled Trial. J Clin Oncol. 2023 Mar 10;41(8):1541-1552. doi: 10.1200/JCO.22.00046. Epub 2023 Jan 19. PMID 36657089
- [Background] Nerad E, Lahaye MJ, Maas M, Nelemans P, Bakers FC, Beets GL, Beets-Tan RG. Diagnostic Accuracy of CT for Local Staging of Colon Cancer: A Systematic Review and Meta-Analysis. AJR Am J Roentgenol. 2016 Nov;207(5):984-995. doi: 10.2214/AJR.15.15785. Epub 2016 Aug 4. PMID 27490941
- [Background] Brouwer NPM, Stijns RCH, Lemmens VEPP, Nagtegaal ID, Beets-Tan RGH, Futterer JJ, Tanis PJ, Verhoeven RHA, de Wilt JHW. Clinical lymph node staging in colorectal cancer; a flip of the coin? Eur J Surg Oncol. 2018 Aug;44(8):1241-1246. doi: 10.1016/j.ejso.2018.04.008. Epub 2018 Apr 17. PMID 29739638
- [Background] van den Beukel BAW, Stommel MWJ, van Leuven S, Strik C, IJsseldijk MA, Joosten F, van Goor H, Ten Broek RPG. A Shared Decision Approach to Chronic Abdominal Pain Based on Cine-MRI: A Prospective Cohort Study. Am J Gastroenterol. 2018 Aug;113(8):1229-1237. doi: 10.1038/s41395-018-0158-9. Epub 2018 Jun 27. PMID 29946174